CLINICAL TRIAL: NCT04748965
Title: Imaging-Guided Vessel Sizing in the Tibial Arteries
Acronym: iVEST
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY20210833
Record Dates: First submitted 2020-12-12; First posted 2021-02-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Artery Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia | interventions — Angiography, Digital Subtraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tibial Vessel Involvement in Patients with peripheral artery disease and CLI: The primary goal is to establish a protocol for performing optimal OCT in below-the-knee vessels. OCT images will be analyzed for lesion characteristics, lesion sizing pre- and post-intervention. This will be analyzed against QVA and IVUS (latter if applicable).
  Interventions: Diagnostic Test: Digital Subtraction Angiography

INTERVENTIONS:
Diagnostic Test: Digital Subtraction Angiography — Compare optical coherence tomography lesion sizing and characteristics compared to traditional digital subtraction angiography

SUMMARY:
This study aims to investigate the utilization of intravascular imaging in treatment of tibial vessels in peripheral artery disease and critical limb ischemia (CLI). The primary goal is to compare optical coherence tomography (OCT) with traditional digital subtraction angiography (DSA) in determining best treatment strategy and vessel optimization, in an effort to improve long term patency and successful wound healing in CLI. Secondary comparison with intravascular ultrasound (IVUS) is undertaken when clinically feasible. The hypothesis is that the adjunctive use of intravascular imaging will affect vessel sizing and anticipated treatment modalities, and therein affect the long term primary patency rates.

DETAILED DESCRIPTION:
This is a prospective, nonrandomized trial to investigate the adjunctive use of intravascular imaging in tibial vessel interventions. The evaluation of OCT is primarily to: (a) establish feasibility and reproducibility in below-the-knee vessels, (b) determine the optimal protocol imaging to produce the optimal clear image frame and clear image length, (c) provide detailed lesion characteristics of tibial disease, (d) assess for luminal gain post-intervention. Operator-determined sizing will be compared against University Hospitals Core Imaging Laboratory assessment of OCT, IVUS (when applicable), and quantitative vessel analysis (QVA).

Subjects will follow up per routine care with corresponding ankle-brachial index and toe-brachial index at 1, 3, 6, and 12 months or as clinically indicated. Wound and amputation data will be collected at the pre-procedural visit and with each subsequent visit. Wound care will be managed by our wound care associates in podiatry, vascular medicine, vascular surgery, or plastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patients with presence of Rutherford IV-VI
* Presence of ≥1 tibial artery involvement requiring endovascular treatment

Exclusion Criteria:

* Patients who do not have tibial disease appropriate for intervention
* Estimated glomerular filtration rate <30 mL/min not on hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tibial vessel involvement in patients with underlying peripheral artery disease and critical limb ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-06-09 (Actual); Study Completion 2024-06-09 (Actual)

PRIMARY OUTCOMES:
Standardized Technique for OCT Use in the Lower Limb | 12 months
  To develop a protocolized, reproducible technique to maximize the Clear Image Length (CIL) on 75 mm pullbacks using 100% contrast in the tibial arteries. The goal is to compare intravascular ultrasound (IVUS) and optical coherence tomography (OCT) with traditional digital subtraction angiography (DSA) in determining best treatment strategy and vessel optimization, in an effort to improve long term patency and successful wound healing in CLI. The hypothesis is that the adjunctive use of intravascular imaging will affect vessel sizing and anticipated treatment modalities, and therein affect the long term primary patency rates.

SECONDARY OUTCOMES:
Comparison of Percent Contrast | 12 months
  CIL in 100% contrast versus 50% contrast/heparinized saline mixture
Vessel Characteristics: Minimal Lumen Area | 12 months
  minimal lumen area (mm^2)
Vessel Characteristics: Reference Vessel Diameter | 12 months
  reference vessel diameter (mm)
Vessel Characteristics: Reference Vessel Area | 12 months
  reference vessel area (mm^2)
Vessel Characteristics: Percentage Stenosis | 12 months
  percentage stenosis (%) on pre-intervention imaging
Plaque Characteristics: Morphology | 12 months
  Percentage composition of calcium, fibrous, or lipid plaque (%)
Plaque Characteristics: Calcium Arc | 12 months
  Calcium arc (degree)
Plaque Characteristics: Calcium Depth | 12 months
  depth of calcium (micron)
Plaque Characteristics: Fibrous cap | 12 months
  depth of fibrous cap (micron)
Attenuation | 12 months
  Measurement of attenuation coefficient (μ OCT) to quantify the strength of interaction of light and tissue
Vessel Characteristics Following Intervention: Luminal Gain | 12 months
  Post-intervention luminal gain (%), plaque modification, and dissections
Vessel Characteristics Following Intervention: Plaque Modification | 12 months
  Reduction in calcium depth (%) if atherectomy is performed
Vessel Characteristics Following Intervention: Dissections | 12 months
  Qualitative description of dissections seen on post-intervention imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (3):
- United States (3):
  - University Hospitals Ahuja Medical Center, Beachwood, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezerra HG, Attizzani GF, Sirbu V, Musumeci G, Lortkipanidze N, Fujino Y, Wang W, Nakamura S, Erglis A, Guagliumi G, Costa MA. Optical coherence tomography versus intravascular ultrasound to evaluate coronary artery disease and percutaneous coronary intervention. JACC Cardiovasc Interv. 2013 Mar;6(3):228-36. doi: 10.1016/j.jcin.2012.09.017. PMID 23517833
- [Background] Witzenbichler B, Maehara A, Weisz G, Neumann FJ, Rinaldi MJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Brodie BR, Stuckey TD, Mazzaferri EL Jr, Xu K, Parise H, Mehran R, Mintz GS, Stone GW. Relationship between intravascular ultrasound guidance and clinical outcomes after drug-eluting stents: the assessment of dual antiplatelet therapy with drug-eluting stents (ADAPT-DES) study. Circulation. 2014 Jan 28;129(4):463-70. doi: 10.1161/CIRCULATIONAHA.113.003942. Epub 2013 Nov 26. PMID 24281330
- [Background] Wijns W, Shite J, Jones MR, Lee SW, Price MJ, Fabbiocchi F, Barbato E, Akasaka T, Bezerra H, Holmes D. Optical coherence tomography imaging during percutaneous coronary intervention impacts physician decision-making: ILUMIEN I study. Eur Heart J. 2015 Dec 14;36(47):3346-55. doi: 10.1093/eurheartj/ehv367. Epub 2015 Aug 4. PMID 26242713
- [Background] Scoccianti M, Verbin CS, Kopchok GE, Back MR, Donayre CE, Sinow RM, White RA. Intravascular ultrasound guidance for peripheral vascular interventions. J Endovasc Surg. 1994 Sep;1:71-80. doi: 10.1583/1074-6218(1994)0012.0.CO;2. PMID 9234107
- [Background] Arthurs ZM, Bishop PD, Feiten LE, Eagleton MJ, Clair DG, Kashyap VS. Evaluation of peripheral atherosclerosis: a comparative analysis of angiography and intravascular ultrasound imaging. J Vasc Surg. 2010 Apr;51(4):933-8; discussion 939. doi: 10.1016/j.jvs.2009.11.034. Epub 2010 Jan 15. PMID 20080002
- [Background] Secco GG, Grattoni C, Parisi R, Oshoala K, Cremonesi A, Fattori R, Castriota F. Optical Coherence Tomography Guidance during Peripheral Vascular Intervention. Cardiovasc Intervent Radiol. 2015 Jun;38(3):768-72. doi: 10.1007/s00270-014-0868-3. Epub 2014 Mar 5. No abstract available. PMID 24595662
- [Background] Eberhardt KM, Treitl M, Boesenecker K, Maxien D, Reiser M, Rieger J. Prospective evaluation of optical coherence tomography in lower limb arteries compared with intravascular ultrasound. J Vasc Interv Radiol. 2013 Oct;24(10):1499-508. doi: 10.1016/j.jvir.2013.06.015. Epub 2013 Aug 17. PMID 23962439
- [Background] Paraskevopoulos I, Spiliopoulos S, Davlouros P, Karnabatidis D, Katsanos K, Alexopoulos D, Siablis D. Evaluation of below-the-knee drug-eluting stents with frequency-domain optical coherence tomography: neointimal hyperplasia and neoatherosclerosis. J Endovasc Ther. 2013 Feb;20(1):80-93. doi: 10.1583/12-4091.1. PMID 23391087
- [Background] Agarwal S, Sud K, Shishehbor MH. Nationwide Trends of Hospital Admission and Outcomes Among Critical Limb Ischemia Patients: From 2003-2011. J Am Coll Cardiol. 2016 Apr 26;67(16):1901-13. doi: 10.1016/j.jacc.2016.02.040. Epub 2016 Mar 21. PMID 27012780
- [Background] Ferraresi R, Mauri G, Losurdo F, Troisi N, Brancaccio D, Caravaggi C, Neri L. BAD transmission and SAD distribution: a new scenario for critical limb ischemia. J Cardiovasc Surg (Torino). 2018 Oct;59(5):655-664. doi: 10.23736/S0021-9509.18.10572-6. Epub 2018 May 22. PMID 29786411